CLINICAL TRIAL: NCT06219746
Title: 99mTc-MIP-1404 SPECT/CT for Primary PROstate Cancer STAging: Comparative Prospective, Randomized Trial to Present Guideline Imaging
Brief Title: 99mTc-MIP-1404 SPECT/CT in Primary Staging of Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Otto Ettala, Adjunct professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: T19/2021
Record Dates: First submitted 2023-11-03; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: PSMA; PET; SPECT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Subjects undergo bone scintigraphy and whole body CT
- Experimental arm (Experimental): Subjects undergo bone scintigraphy, whole body CT, 99mTc-MIP-1404 SPECT/CT, and 18F- PSMA-1007 PET/CT
  Interventions: Diagnostic Test: PSMA-imaging

INTERVENTIONS:
Diagnostic Test: PSMA-imaging — Subjects undergo additional imaging i.e. PSMA/SPECT/CT and PSMA/PET/CT
  Arms: Experimental arm

SUMMARY:
Prostate cancer (PCa) is currently the most common cancer in men in Finland (www.cancerregistry.fi). Although prognosis is very good in majority of men, it is noteworthy that still up to 20% of PCa cases are metastatic at the time of initial diagnosis and yearly 900 men die because of prostate cancer. Robust primary staging is, therefore, one of the most important prognostic factors, and it is crucial for treatment decision. Despite their low sensitivity to detect metastasis, bone scintigraphy (BS) and contrast enhanced whole body computed tomography (ce-wbCT) are recommended by current guidelines for primary staging in men at risk of metastasis.

MIP-1404 is a small-molecule PSMA inhibitor that can be used in SPECT systems (99mTc-MIP- 1404 SPECT/CT). 99mTc-MIP-1404 SPECT/CT is performed by a single IV bolus of 99mTc-MIP-1404, which binds with high affinity to extracellular domain of PSMA molecule. As of March 2020, a total of 629 subjects have received 99mTc-MIP-1404 injection averaging 740 ±111 MBq (20 ± 3 mCi) per administration in prospective clinical trials. 99mTc MIP-1404 has been well tolerated following a single IV dose at 740 ± 111 MBq in both healthy volunteers and patients with confirmed metastatic prostate adenocarcinoma. In prospective and retrospective studies, it has shown high potential to detect prostate cancer lesions in primary staging. In fact, Goffin et al. reported a sensitivity of 50% and specificity of 87% detecting local lymph node metastasis in radically operated patients when histopathology was used as a reference. This corresponds closely to the sensitivity of PSMA-PET.

PROSTAMIP is a randomized prospective single-institutional study to demonstrate superiority of 99mTc-MIP-1404 SPECT/CT compared to traditional imaging modalities (99mTc-HMDP planar BS plus ce-wbCT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol
* Subjects must be male, aged 18 years or above at Baseline
* Histopathologically confirmed high risk (Gleason ≥4+4, PSA ≥20 and/ or cT≥3a) acinar or ductal adenocarcinoma of prostate

Exclusion Criteria:

* Allergy/sensitivity to study medications or their ingredients
* Subjects unable to provide written informed consent
* Subjects who have any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk by participation in the study, or may influence the result of the study.
* Subjects who have a history of drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Subjects who have androgen deprivation therapy initiated before enrolment
* Subjects who have claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with local lymph node metastasi(e)s | Baseline
  Superiority of experimental arm (99mTc-MIP-1404 SPECT/CT) in detecting subjects with local lymph node metastasi(e)s compared to control arm (ce-wbCT)

SECONDARY OUTCOMES:
Number of subjects with metastasis | Baseline
  Comparison of detection of metastatic subjects (local lymph node metastasis and/ or distant metastasis) in experimental arm (99mTc-MIP-1404 SPECT/CT) and in control arm (a combination of 99mTc-HMDP planar bone scintigraphy and contract enhanced CT)
Diagnostic accuracy of detecting subjects with metastasis between PSMA-SPECT/CT and conventional imaging | Baseline
  Comparison of diagnostic accuracy between PSMA-SPECT/CT and conventional imaging (a combination of 99mTc-HMDP planar BS and ce-wbCT) in detection of metastatic subjects (a combination of nodal and distant metastasis)
True positive rate in lesion level between PSMA-SPECT/CT and conventional imaging | Baseline
  Description of true positive rate of metastatic lesions between PSMA-SPECT/CT and conventional imaging (a combination of 99mTc-HMDP planar bone scintigraphy and contrast enhanced)
False positive rate in lesion level between PSMA-SPECT/CT and conventional imaging | Baseline
  Description of false positive rate of metastatic lesions between PSMA-SPECT/CT and conventional imaging (a combination of 99mTc-HMDP planar bone scintigraphy and contrast enhanced)
False negative rate in lesion level between PSMA-SPECT/CT and conventional imaging | Baseline
  Description of false negative rate of metastatic lesions between PSMA-SPECT/CT and conventional imaging (a combination of 99mTc-HMDP planar bone scintigraphy and contrast enhanced)
Diagnostic accuracy of detecting subjects with metastasis between PSMA-SPECT/CT and PSMA-PET/CT | Baseline
  Comparison of diagnostic accuracy between PSMA-SPECT/CT and PSMA-PET/CT in detection of metastatic subjects (a combination of nodal and distant metastasis)
True positive rate in lesion level between PSMA-SPECT/CT and PSMA-PET/CT | Baseline
  Description of true positive rate of metastatic lesions between PSMA-SPECT/CT and PSMA-PET/CT
False positive rate in lesion level between PSMA-SPECT/CT and PSMA-PET/CT | Baseline
  Description of false positive rate of metastatic lesions between PSMA-SPECT/CT and PSMA-PET/CT
False negative rate in lesion level between PSMA-SPECT/CT and PSMA-PET/CT | Baseline
  Description of false negative rate of metastatic lesions between PSMA-SPECT/CT and PSMA-PET/CT
Inter-rater agreement | Baseline
  Cohen´s Kappa value between the two readers in each imaging modality
Effect on treatment decision | Baseline
  The number and proportion of subjects in which treatment recommendation was changed due to 99mTc-MIP 1404 SPECT/CT or 18F-PSMA-1007 PET/CT

OTHER OUTCOMES:
PSMA only lesions | Baseline
  Characterization of PSMA only lesions
ctDNA | Baseline
  Comparison ctDNA between non-metastatic patients, patients with PSMA only lesions and patients with lesions seen in conventional imaging
Gut microbiota | Baseline
  Comparison results of shotgun metagenomic analysis of gut microbiota between non-metastatic patients, patients with PSMA only lesions and patients with lesions seen in conventional imaging
Optimization of 99mTc-MIP-1404 SPECT/CT imaging protocol | Baseline
  The shortest acquisition time with acceptable decrease in diagnostic accuracy of detecting local lymph node metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Otto O Ettala, Principal Investigator — Turku University Hospital
Locations (1):
- University Hospital of Turku, Hospital Distric of Southwest Finland, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No